CLINICAL TRIAL: NCT00567060
Title: A Multicenter, Randomized, Double Blind, Placebo Controlled, Parallel Group Study of the Efficacy and Safety of 9600 and 4800 mg/Day Piracetam Taken for 12 Months by Subjects Suffering From Mild Cognitive Impairment (MCI)
Brief Title: Efficacy and Safety of Piracetam Taken for 12 Months in Subjects Suffering From Mild Cognitive Impairment (MCI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N01001
Record Dates: First submitted 2007-11-30; First posted 2007-12-04 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2009-09

CONDITIONS: Memory Disorders
Keywords: Piracetam; Nootropil
MeSH Terms: conditions — Memory Disorders | interventions — Piracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Piracetam

SUMMARY:
The purpose of this study was to explore in a more documented way the relative potential and efficacy of piracetam 9600 and 4800 mg daily.

ELIGIBILITY:
Inclusion Criteria:

* male/female between 50 and 89 years (inclusive)
* declining cognitive function of at least 3 months duration interfering with complex activities of daily living
* normal basic activities of daily independent living
* Clinical Dementia Rating scale score equal to 0.5
* score at least one point above the lowest possible score on 7 out of 8 tests in the cognitive battery at both Selection Visit and Baseline Visit

Exclusion Criteria:

* general anesthetics within 3 months of selection visit
* history of severe allergic drug reaction(s)
* history of drug or alcohol dependence (DSM IV defined) within the last 12 months
* any drug prescribed to activate cerebral metabolism, taken within 1 week of screening or/and concomitantly
* concomitant intake of anticoagulent medications
* concomitant intake or intake within 1 week before screening of drug that might affect cognitive function or central nervous system
* history of dementia, psychiatric or neurological disorders, mental retardation, learning disabilities and stroke
* current depression
* impaired renal function, thyroid function or neurological degeneration
* any gastrointestinal dysfunction that might interfere with the absorption or elimination of the study drug
* insulin-dependant diabetes mellitus
* bleeding disorders or disturbance in hemostatic function.

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 676 (Actual)
Dates: Start 2000-05; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Cognitive Battery Composite Score over a 52-week period

SECONDARY OUTCOMES:
safety of piracetam for 12 months

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma

REFERENCES:
- [Result] Jelic V, Kivipelto M, Winblad B. Clinical trials in mild cognitive impairment: lessons for the future. J Neurol Neurosurg Psychiatry. 2006 Apr;77(4):429-38. doi: 10.1136/jnnp.2005.072926. Epub 2005 Nov 23. PMID 16306154